CLINICAL TRIAL: NCT06706466
Title: Systemic Immune-Inflammation Index As a Predictor of Neoadjuvant Treatment Efficacy in Advanced Gastric Cancer Based on a Dynamic Clinical Model
Brief Title: Evaluate the Prognostic Significance of Changes in the Systemic Immune-Inflammation Index in Patients with AGC Treated with ICI Therapy.
Status: Completed | Type: Observational
Sponsor: Chang-Ming Huang, Prof. (Other)
Responsible Party: Sponsor-Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: 2024KY247
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Immunotherapy Gastrict Cancer; Inflammation Biomarkers; Gastric Cancers
Keywords: Inflammation Index; gastric cancer; immunotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SIIR-Dec: Patients with an SIIR of ≥-0.3 after ICI treatment
  Interventions: Other: observational study
- SIIR-non-Dec: Patients with an SIIR of < -0.3 after ICI treatment
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — Non-interventional

SUMMARY:
The SIIR during neoadjuvant therapy can serve as a specific biomarker for predicting the efficacy of immunotherapy in patients with advanced gastric cancer.

DETAILED DESCRIPTION:
A total of 410 patients with advanced gastric cancer treated with neoadjuvant chemotherapy (NAC group, 178) or immunotherapy (ICIs group, 232) were enrolled in two tertiary referral centers. The SIIR ([SIIpost-treatment - SIIpre-treatment] / SIIpre-treatment) was calculated. The diagnostic threshold for SIIR was set at the median value (-0.3) A joint model based on longitudinal trajectory and time-to-event analysis was used to assess the correlation between SIIR and the risk of death in patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

(1) preoperative clinical staging of cT2-4NxM0; (2) primary gastric adenocarcinoma confirmed via pathology; (3) no distant metastasis to the liver, lungs, or abdominal cavity as confirmed through preoperative chest X-ray or chest CT, abdominal ultrasound, and abdominal CT; (4) All patients received neoadjuvant therapy, followed by gastrectomy.

Exclusion Criteria:

We excluded patients under 18 or over 80, those with distant metastasis, remnant gastric cancer, prior radiotherapy, other malignancies, abdominal surgery history (except laparoscopic cholecystectomy), recent unstable angina, myocardial infarction, cerebrovascular accidents, or those requiring emergency surgery due to disease progression

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective analysis included 453 patients diagnosed with advanced gastric adenocarcinoma (T2-4aNx/+M0, according to the 7th edition of the American Joint Committee on Cancer [18]) who received treatment between January 2018 and December 2021. Finally, 410 patients met the inclusion criteria. Ethical approval for this study.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
survival | 36 months
  Telephone follow-up

SECONDARY OUTCOMES:
recurrence | 36 months
  Telephone follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No